CLINICAL TRIAL: NCT01173991
Title: Clinical Assessment of Carbohydrate Counting in Adult Patients With Type 1 Diabetes Treated With Continuous Subcutaneous Insulin Infusion: a Randomized Controlled Study (GIOCAR)
Brief Title: Carbohydrate Counting in Adults With Type 1 Diabetes Treated With Continuous Subcutaneous Insulin Infusion
Acronym: GIOCAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Emanuele Bosi, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIOCAR
Record Dates: First submitted 2010-07-26; First posted 2010-08-03 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus, Type 1; Insulin Pump, Programmable
Keywords: carbohydrate counting; continuous subcutaneous insulin infusion; type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbohydrate counting (Experimental): This group received carbohydrate counting training
  Interventions: Behavioral: Carbohydrate counting training
- Controls (No Intervention): This group received standard education
  Interventions: Behavioral: Carbohydrate counting training

INTERVENTIONS:
Behavioral: Carbohydrate counting training — Carbohydrate counting was taught during 4-5 individual sessions with a dietician and a diabetologist.

SUMMARY:
The investigators postulate that carbohydrate (CHO) counting in adult patients with type 1 diabetes mellitus (T1DM) treated with continuous subcutaneous insulin infusion (CSII) may improve glycemic control, glycemic variability and quality of life.

DETAILED DESCRIPTION:
This study was designed as a randomized, controlled (versus standard education), open, one-center trial. Patients in group 1 were taught carbohydrate counting to estimate insulin preprandial bolus, while the patients in group 2 followed standard education. Primary outcome (glycosylated hemoglobin, HbA1c) and secondary outcomes (fasting glucose, glycemic variability, insulin requirement, body mass index (BMI), waist circumference, quality of life) were measured at baseline, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes mellitus
* age 18-65
* continuous subcutaneous insulin infusion for at least 3 months

Exclusion Criteria:

* patients who have already been trained in carbohydrate counting
* known hypothyroidism not on replacement therapy
* renal disease (serum creatinine >1.4 mg/dl in females and >1.7 mg/dl in males)
* patients with celiac disease
* pregnancy
* serious diseases or disabilities which may interfere with study assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) | 6 months

SECONDARY OUTCOMES:
Fasting glucose | 6 months
Glycemic variability (mean, sd, min, max, variability range, BG in target range, LBGI, HBGI) based on capillary glucose data | 6 months
Daily insulin requirement (basal daily requirement, bolus daily requirement, total daily requirement) | 6 months
Body Mass Index (BMI) | 6 months
Waist circumference | 6 months
Quality of life by Diabetes Specific Quality of Life Scale (DSQOLS) questionnaire | 6 months
Hypoglycemia (capillary glucose<50 mg/dl) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Bosi, MD, Principal Investigator — San Raffaele Scientific Institute, Milano Italy
Locations (1):
- San Raffaele Scientific Institute, Milan, Italy